CLINICAL TRIAL: NCT01641185
Title: Hypofractionated Ion Irradiation (Carbon Ions Versus Protons) of the Prostate
Brief Title: Ion Prostate Irradiation
Acronym: IPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Prof. Dr. Herfarth, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Neoplasms
Keywords: prostate; IPI; hypofractionation; carbon ions; proton
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- protons (Experimental): irradiation 20 x 3,3 GyE protons
  Interventions: Procedure: radiation
- carbon ions (Experimental): irradiation 20 x 3,3 GyE carbon ions
  Interventions: Procedure: radiation

INTERVENTIONS:
Procedure: radiation — radiation with protons or carbon ions

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of primary hypofractionated irradiation of the prostate with carbon ions or protons using the raster scan technique.

DETAILED DESCRIPTION:
as published: Habl G, Hatiboglu G, Edler L, Uhl M, Krause S, Roethke M, Schlemmer HP, Hadaschik B, Debus J, Herfarth K: Ion Prostate Irradiation (IPI) - a pilot study to establish the safety and feasibility of primary hypofractionated irradiation of the prostate with protons and carbon ions in a raster scan technique. BMC cancer 2014, 14(1):202.

http://www.ncbi.nlm.nih.gov/pubmed/24641841

ELIGIBILITY:
Inclusion Criteria:

histological proven carcinoma of the prostate with Gleason score risk of lymphe node involvement of <15% calculated by the Yale-formula; Risk [%] = [GS -5] x [PSA/3 + 1.5 x T], mit T = 0, 1, and 2 for cT1c, cT2a, und cT2b/cT2c

* Karnofsky-Index ≥ 70%
* age between 40 and 80 years
* PSA

Exclusion Criteria:

Stadium IV (distant metastases) Lymphogenous Metastases hip replacement former irradiation of the pelvis pacemaker defibrillator

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
proctitis and cystitis | 3 years
  via incidence grade 3-4 toxicity (NCI-CTC-AE)

SECONDARY OUTCOMES:
PSA-PFS | 3 years
  by measuring PSA values every 3 months
OS | 3 years
quality of life | 3 years
  by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, Prof. Dr., Principal Investigator — University Hospital of Heidelberg
Locations (1):
- University of Heidelberg, Radiooncology, HIT, Heidelberg, Germany

REFERENCES:
- [Background] Habl G, Hatiboglu G, Edler L, Uhl M, Krause S, Roethke M, Schlemmer HP, Hadaschik B, Debus J, Herfarth K. Ion Prostate Irradiation (IPI) - a pilot study to establish the safety and feasibility of primary hypofractionated irradiation of the prostate with protons and carbon ions in a raster scan technique. BMC Cancer. 2014 Mar 19;14:202. doi: 10.1186/1471-2407-14-202. PMID 24641841
- [Background] Habl G, Uhl M, Katayama S, Kessel KA, Hatiboglu G, Hadaschik B, Edler L, Tichy D, Ellerbrock M, Haberer T, Wolf MB, Schlemmer HP, Debus J, Herfarth K. Acute Toxicity and Quality of Life in Patients With Prostate Cancer Treated With Protons or Carbon Ions in a Prospective Randomized Phase II Study--The IPI Trial. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):435-443. doi: 10.1016/j.ijrobp.2016.02.025. Epub 2016 Feb 12. PMID 27084659